CLINICAL TRIAL: NCT02227576
Title: Secondary Prophylaxis Use of Romiplostim for the Prevention of Thrombocytopenia Induced by Temozolomide in Newly Diagnosed Glioblastoma Patients
Brief Title: Prevention of Thrombocytopenia in Glioblastoma Patients
Acronym: PLATUM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted for efficacy following the results of the interim analysis provided for in the protocol on 20 patients.
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011_29; 2012-001751-38 (EudraCT Number)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Thrombocytopenia; Glioblastoma
Keywords: glioblastoma, thrombocytopenia, temozolomide, chemotherapy
MeSH Terms: conditions — Thrombocytopenia; Glioblastoma | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Romiplostim (Experimental): Romiplostim lyophilized formulation is a white, solide cake that is reconstituted with sterile water for injection.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim

SUMMARY:
Chemotherapy used in the treatment of primitive tumors of the central nervous system has a particularly important platelet toxicity compared to chemotherapy used for treatment of other tumors. Chemotherapy postponed for toxicity is often due to thrombocytopenia (TP). The TP and/or the other anomalies of coagulation, which can be spontaneous (Rogers, 2004) or induced (Gerber, 2006) can have dramatic consequences:

* specifically neurological (intratumoral bleeding with particularly important neovascularization) with a functional aggravation and sometimes involvement of vital prognosis,
* digestive (Garcia-Rodiguez, 2001) in patients receiving long term treatment with corticoids (potential gastric toxicity).

The encouraging results from the EORTC/NCIC trial by Stupp (median survival among patients with newly diagnosed glioblastoma is 14.6 months with an estimated 5-year survival of 9, 8%), has changed the standard of care of these patients (Stupp et al., 2009). Patients with newly diagnosed, histologically confirmed glioblastoma receive radiotherapy (2 Gy given 5 days per week for 6 weeks, for a total of 60 Gy) plus continuous daily Temozolomide (75 mg per square meter of body-surface area per day, 7 days per week from the first to the last day of radiotherapy), followed by six cycles of adjuvant Temozolomide (TMZ) (150 to 200 mg per square meter for 5 days during each 28-day cycle). The Stupp regimen is currently the treatment of reference for glioblastoma and is used as a basis in various clinical studies with new agents.

This study aims to evaluate Romiplostim for the treatment of TP secondary to initial TMZ chemotherapy of glioblastomas.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of newly diagnosed glioblastoma,
* Age: 18 and older,
* Information to patient and signed consent form,
* Indication for a " Stupp " protocol (cerebral focal radiotherapy and concomitant TMZ followed by adjuvant TMZ - 6 cycles),
* Patient with grade 3 or 4 TP during Temozolomide chemotherapy, regardless of when the onset of TP was: after completion of concomitant RT/CT, before adjuvant CT or during adjuvant CT and only if a minimum of 2 cycles are still planned,
* Normal initial platelets count (> 100 000/mm3) before the start of Temozolomide during the RT/CT concomitant phase,
* Adequate haematological, renal, hepatic function at the time of inclusion visit,
* ECOG PS 0-2 (patients unable to walk because of a paralysis and who are up in a wheel chair will be considered as ambulatory for the evaluation of the ECOG performance status),
* Life expectancy > 2 months,
* Patients covered by the French Health Insurance System,
* Negative pregnancy test at the time of inclusion visit,
* If required, effective contraception respecting criteria of CPMP/ICH/286/95 (such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner).

Exclusion Criteria:

* Concomitant radiotherapy (Romiplostim will be started after the completion of the RT/CT concomitant phase),
* Other malignancies (prior hx malignancies),
* Any anterior systemic chemotherapy,
* Any known coagulation disease or known haematological disease even if resolved. Known hypercoagulate state (e.g., factor V Leiden, protein C defiency, protein S deficiency, PT 20201, antiphospholipid antibody syndrome…),
* Prior Romiplostim exposure or prior exposure to other TPO mimetics,
* History of thromboembolic disease < 6 months. Treatment with anticoagulant such as Heparin or antivitamin K (LMWH as prophylactic treatment is authorized),
* Any other hemato-toxicity (anemia, neutropenia) requiring EPO or GCSF,
* Other causes of Temozolomide interruption (non haematological toxicities),
* Known hypersensitivity to any E-coli derived product,
* Participation to any other study during the last 30 days,
* Refusal to give written informed consent,
* Pregnancy or nursing,
* For all men and women of childbearing potential: Refusal or inability to use effective means of contraception,
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial,
* Persons protected by a legal regime (guardianship, trusteeship),
* Patients in emergency situations,
* Patients kept in detention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving 100% of the planned TMZ dosage in the whole Stupp protocol. The primary endpoint will consider dose reduction and dose delay. | one year

SECONDARY OUTCOMES:
Incidence of serious adverse events according to CTCAE 4.0 criteria. | one year
Incidence of delayed chemotherapy cycles and the incidence of chemotherapy cycles with dose reduction due to severe TP | one year
Number and percentage of patients with TP of grade 3 or grade 4 after receiving Romiplostim. | One year
Number and percentage of patients receiving platelets transfusion for TP | one year
Incidence and type of adverse events linked to TP episodes during Romiplostim and Temozolomide combined treatment. | one year
6 months Progression Free Survival: | one year

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Le Rhun, MD, Principal Investigator — CHRU LILLE
Locations (4):
- France (4):
  - CHRU de Lille, Hôpital Roger Salengro,Clinique de Neurochirurgie, Lille
  - Hôpital Neurologique Pierre Wertheimer, Lyon,, Lyon
  - AP-HM,Hôpital La Timone, AP-HM, Marseille, Marseille
  - AH-HP, Hôpital Pitié-Salpêtrière, Service de Neurologie 2, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong TS, Cao Y, Scheurer ME, Vera-Bolanos E, Manning R, Okcu MF, Bondy M, Zhou R, Gilbert MR. Risk analysis of severe myelotoxicity with temozolomide: the effects of clinical and genetic factors. Neuro Oncol. 2009 Dec;11(6):825-32. doi: 10.1215/15228517-2008-120. PMID 19179423
- [Background] Gerber DE, Grossman SA, Zeltzman M, Parisi MA, Kleinberg L. The impact of thrombocytopenia from temozolomide and radiation in newly diagnosed adults with high-grade gliomas. Neuro Oncol. 2007 Jan;9(1):47-52. doi: 10.1215/15228517-2006-024. Epub 2006 Nov 15. PMID 17108062
- [Background] George JN, Raskob GE, Shah SR, Rizvi MA, Hamilton SA, Osborne S, Vondracek T. Drug-induced thrombocytopenia: a systematic review of published case reports. Ann Intern Med. 1998 Dec 1;129(11):886-90. doi: 10.7326/0003-4819-129-11_part_1-199812010-00009. PMID 9867731
- [Background] Kuter DJ, Rummel M, Boccia R, Macik BG, Pabinger I, Selleslag D, Rodeghiero F, Chong BH, Wang X, Berger DP. Romiplostim or standard of care in patients with immune thrombocytopenia. N Engl J Med. 2010 Nov 11;363(20):1889-99. doi: 10.1056/NEJMoa1002625. PMID 21067381
- [Background] Molineux G. The development of romiplostim for patients with immune thrombocytopenia. Ann N Y Acad Sci. 2011 Mar;1222:55-63. doi: 10.1111/j.1749-6632.2011.05975.x. PMID 21434943
- [Background] Sure D, Dunn I, Norden A, Anderson WS. Intracerebral hemorrhage secondary to thrombocytopenia in a patient treated with temozolomide. Clin Neurol Neurosurg. 2010 Oct;112(8):741-2. doi: 10.1016/j.clineuro.2010.04.005. PMID 20434832
- [Background] Mutter N, Stupp R. Temozolomide: a milestone in neuro-oncology and beyond? Expert Rev Anticancer Ther. 2006 Aug;6(8):1187-204. doi: 10.1586/14737140.6.8.1187. PMID 16925485
- [Background] Oh J, Kutas GJ, Davey P, Morrison M, Perry JR. Aplastic anemia with concurrent temozolomide treatment in a patient with glioblastoma multiforme. Curr Oncol. 2010 Aug;17(4):124-6. doi: 10.3747/co.v17i4.526. PMID 20697524
- [Derived] Le Rhun E, Devos P, Houillier C, Cartalat S, Chinot O, Di Stefano AL, Lepage C, Reyns N, Dubois F, Weller M. Romiplostim for temozolomide-induced thrombocytopenia in glioblastoma: The PLATUM trial. Neurology. 2019 Nov 5;93(19):e1799-e1806. doi: 10.1212/WNL.0000000000008440. Epub 2019 Oct 4. PMID 31586022